CLINICAL TRIAL: NCT02324244
Title: A Prospective Monitoring Study of Cytomegalovirus Infection in Immunocompetent Critical Heart Surgery Patients
Brief Title: CMV Intensive Care Units
Status: Completed | Type: Observational
Sponsor: Emilio Bouza (Other)
Responsible Party: Sponsor-Investigator, Emilio Bouza, Head of Department, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: MICRO.HGUGM.2014-006
Record Dates: First submitted 2014-11-26; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: CMV Infection
Keywords: Cytomegalovirus; critical patient; ICU; immunocompetent; clinical suspicion; risk factors
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- immunocompetent patients underwent heart surgery

SUMMARY:
Prospectively assessment of CMV viremia by real-time polymerase chain reaction (PCR) in a broad cohort of consecutive immunocompetent adults admitted to a major heart surgery intensive care unit (MHS-ICU) with the goal of determining the epidemiology, risk factors, and clinical significance of CMV infection.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Age of at least 18 years
* Admission to the MHS-ICU for at least 72 hours

Exclusion Criteria:

* Inability to give informed consent
* Age younger than 18 years
* AIDS
* Pregnancy
* Organ or bone marrow transplant, receipt of immunosuppressive therapy including corticosteroids within 30 days, and cancer or hematologic malignancy treated with radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: immunocompetent adults admitted to a major heart surgery intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
incidence number of participants with a positive CMV positive result | month 8

SECONDARY OUTCOMES:
risk factors for CMV reactivation | month 8
mortality by day 30 | month 8
  composite endpoint. hospitalization or death by day 30
prolonged hospitalization . More than 30 days | month 8

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Muñoz, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Servicio de Microbiologia y Enfermedades Infecciosas, Madrid, Madrid, Spain